CLINICAL TRIAL: NCT03029234
Title: An Open-label, Single-arm, Phase 3 Study of Carfilzomib in Combination With Dexamethasone in Subjects With Relapsed and Refractory Multiple Myeloma in China
Brief Title: Carfilzomib in Combination With Dexamethasone (Kd) in Chinese Patients With Relapsed & Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140242; CFZ005 (Other: Onyx Therapeutics Inc.)
Record Dates: First submitted 2016-11-11; First posted 2017-01-24 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Dexamethasone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Carfilzomib with Dexamethasone (Experimental): Participants will receive carfilzomib administered by intravenous (IV) infusion on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle (20 mg/m² on days 1 and 2 of cycle 1 and 27 mg/m² thereafter).
  Participants will also receive 20 mg dexamethasone IV or orally on days 1, 2, 8, 9, 15, 16, 22, and 23 of each cycle.
  Participants will receive treatment until disease progression, unacceptable toxicity, initiation of new antimyeloma therapy, withdrawal of consent, non-compliance, or intercurrent illness or worsening of a chronic condition, whichever occurs first.
  Interventions: Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Dexamethasone — 20 mg intravenous (IV) or oral dexamethasone on days 1, 2, 8, 9, 15, 16, 22, and 23 in 28-day cycles.
Drug: Carfilzomib — Infusion of IV carfilzomib on days 1, 2, 8, 9, 15 and 16 in each 28-day cycle.
  Other Names: Kyprolis

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and overall response rate of carfilzomib in combination with dexamethasone for the treatment of multiple myeloma in China.

ELIGIBILITY:
Inclusion Criteria: - Multiple myeloma - Subjects must have measurable disease, defined as one or more of the following: -- Serum M-protein ≥ 1 g/dL -- Urine M-protein ≥ 200 mg/24 hours -- In subjects without measurable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal κ/λ ratio - Subjects must have been responsive (ie, achieved a minimal response [MR] or better) to at least one of their prior treatment regimens - Refractory to the most recently received therapy. Refractory disease defined as ≤ 25% response to, or progressing during therapy or within 60 days after completion of therapy - Subjects must have received ≥ 2 prior regimens. Induction therapy and stem cell transplant (± maintenance) will be considered as 1 regimen - Subjects must have received prior treatment with bortezomib and an immunomodulatory drug - Subjects must have received an alkylating agent or anthracycline alone or in combination with other myeloma treatments (this may include high dose melphalan as part of the conditioning regimen prior to a stem cell transplant) - Males and females ≥ 18 years of age - Life expectancy of more than 3 months - Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 - Adequate hepatic function, with bilirubin < 2.0 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 times the ULN - Absolute neutrophil count (ANC) ≥ 1,000/mm³, hemoglobin ≥ 8.0 g/dL, and platelet count ≥ 50,000/mm³ • Subjects should not have received platelet transfusions for at least 1 week prior to obtaining the screening platelet count • Screening ANC should be independent of granulocyte colony stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF) support for ≥ 1 week and pegylated G-CSF for ≥ 2 weeks • Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed; however, most recent RBC transfusion may not have been done within 7 days prior to obtaining screening hemoglobin - Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/min. Calculated CrCl should be performed by using a widely accepted equation (eg, the Cockcroft and Gault equation): ([140 - Age] × Mass [kg] / [72 × Creatinine mg/dL]). Multiply the result by 0.85 if the subject is female. - Left ventricular ejection fraction (LVEF) ≥ 40%; 2-dimensional transthoracic echocardiogram (ECHO) is the preferred method of evaluation; multiple gated acquisition scan (MUGA) is acceptable if ECHO is not available - Written informed consent in accordance with federal, local, and institutional guidelines - Female subjects of child-bearing potential (FCBP) must have a negative serum pregnancy test within 21 days prior to enrollment and agree to use an effective method of contraception during and for 30 days following last dose of carfilzomib. This protocol defines a FCBP as a sexually mature woman who: 1) has not undergone a hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) - Male subjects must use an effective barrier method of contraception during the study and for 3 months following the last dose of carfilzomib if sexually active with a FCBP. Male subjects must not donate sperm during treatment and for an additional 90 days after last dose of carfilzomib. Male subjects with pregnant partners must practice sexual abstinence or use a condom during vaginal sex. Exclusion Criteria: - Waldenström's macroglobulinemia or immunoglobulin M (IgM) multiple myeloma - Subjects who failed to achieve at least a confirmed MR on any of their prior regimens - Subjects with non-secretory multiple myeloma, defined as < 1 g/dL M-protein in serum and < 200 mg/24 hour M-protein in urine and SFLC ≤ 100 mg/L (involved light chain) - Glucocorticoid therapy (prednisone > 10 mg/day or equivalent) within 3 weeks prior to Cycle 1 Day 1 - POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) - Plasma cell leukemia (> 2.0 × 10⁹/L circulating plasma cells by standard differential) - Chemotherapy with approved or investigative anticancer therapeutics including steroid therapy within the 3 weeks prior to Cycle 1 Day 1 - Radiation therapy or immunotherapy in the 4 weeks prior to Cycle 1 Day 1; localized radiation therapy within 1 week prior to Cycle 1 Day 1 - Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (T½) prior to Cycle 1 Day 1, whichever time is greater - Prior treatment with carfilzomib - Major surgery within 3 weeks before Cycle 1 Day 1 - Congestive heart failure (CHF; New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months - Uncontrolled hypertension (a sustained systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg) - Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to Cycle 1 Day 1 - Known human immunodeficiency virus (HIV) seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed) - Non-hematologic malignancy within the past 3 years except: -- Adequately treated basal cell or squamous cell skin cancer, -- Carcinoma in situ of the cervix, or -- Prostate cancer < Gleason Score 6 with stable prostate-specific antigen - Subjects with treatment-related myelodysplastic syndrome - Significant neuropathy (Grade 3, 4, or Grade 2 with pain) at the time of baseline evaluation - Subjects in whom the required program of fluid hydration is contraindicated, eg, due to pre-existing pulmonary, cardiac, or renal impairment - Subjects with known or suspected amyloidosis - Subjects with pleural effusions requiring thoracentesis - Subjects with ascites requiring paracentesis - Any clinically significant medical disease or condition, that in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent - Female subjects who are pregnant or lactating, or planning to become pregnant during treatment and for an additional 30 days after discontinuing carfilzomib. - Serious psychiatric or medical conditions that could interfere with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- China (17):
  - Beijing Chao Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First Peoples Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuang University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Changzheng Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Du J, Fang B, Li J, Jin J, Wang S, Zou D, Cai Z, Wang H, Hu J, Li W, Fu C, Shao Z, Xia Z, Liu P, Niu T, Tang ET, Kimball AS, Hou J, Chen W. A study of carfilzomib and dexamethasone in patients with relapsed and refractory multiple myeloma in China. Int J Hematol. 2021 Mar;113(3):422-429. doi: 10.1007/s12185-020-03044-z. Epub 2021 Jan 3. PMID 33389656
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 18 centers in China. The primary efficacy analysis was prespecified to occur when all enrolled participants had received 6 cycles of therapy or discontinued treatment. This occurred on November 5, 2018. A final analysis for efficacy was prespecified when all enrolled participants had the opportunity to be treated with at least 12 cycles. This occurred on March 15, 2019.
  The final analysis for safety occurred once all participants completed the study, 4 June 2021.
Groups:
- Carfilzomib With Dexamethasone: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle (20 mg/m² on days 1 and 2 of cycle 1 and 27 mg/m² thereafter). Participants also received 20 mg dexamethasone IV or orally on days 1, 2, 8, 9, 15, 16, 22, and 23.
  Participants received treatment until disease progression, unacceptable toxicity, initiation of new antimyeloma therapy, withdrawal of consent, subject noncompliance, or intercurrent illness or worsening of a chronic condition, whichever occurred first.
Period: Overall Study
Arm/Group | Carfilzomib With Dexamethasone
Started | 126
Received Carfilzomib | 123
Completed | 27
Not Completed | 99
Not completed — Sponsor Decision | 1
Not completed — Withdrawal by Subject | 5
Not completed — Death | 91
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all enrolled participants who received at least 1 dose of carfilzomib.
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 123
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 68
    1 (Restricted but ambulatory) | 45
    2 (Ambulatory but unable to work) | 10
Time From Initial Diagnosis to First Dose [Median (Full Range); unit: months] — One participant had a data entry error with year of diagnosis entered as 2017 instead of 2014, leading to an erroneous minimum time since diagnosis reported. Population: Participants with available data
  months
    number analyzed (Participants) | 117
    (all) | 38.70 [0.4 to 182.8]
Total Number of Prior Regimens [Median (Full Range); unit: regimens] | 4.0 [2 to 19]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) After at Least 6 Cycles of Treatment Assessed by the Independent Review Committee
Description: ORR is defined as the percentage of participants with a best overall response of partial response (PR), very good PR (VGPR), complete response (CR), or stringent CR (sCR) based on the International Myeloma Working Group Uniform Response Criteria.
  sCR: As for CR, and absence of clonal plasma cells in bone marrow (BM). CR: No immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and < 5% plasma cells in BM. Normal serum free light chain (SFLC) ratio if disease measurable only by SFLC.
  VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% decrease in serum M-protein with urine M-protein <100 mg/24 hrs. If disease measurable only by SFLC, ≥ 90% decrease in the difference between involved and uninvolved FLC levels (dFLC).
  PR: ≥ 50% reduction of serum M-protein and ≥ 90% reduction in urine M-protein or to < 200 mg/24 hrs, or a ≥ 50% decrease in dFLC. A ≥ 50% decrease in the size of soft tissue plasmacytomas present at baseline.
Time Frame: Response was assessed every 28 days until disease progression; ORR was analyzed after all participants received at least 6 cycles or discontinued treatment; the data cut-off date was 5 November 2018; median follow-up time for progression was 8.9 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 35.8 [27.3 to 44.9]
Statistical Analysis 1: Comparison: Carfilzomib With Dexamethasone; Test type: Other — The prespecified threshold that the primary endpoint would be met was if the lower limit of the 95% confidence interval (CI) was greater than 18%; Overall response rate = 35.8, 95% CI 2-sided [27.3 to 44.9]

2. Secondary Outcome: Overall Response Rate (ORR) After at Least 6 Cycles of Treatment Assessed by the Investigator
Description: as for outcome 1
Time Frame: Response was assessed every 28 days until disease progression; ORR was analyzed after all participants received at least 6 cycles or discontinued treatment; the data cut-off date was 05 November 2018; median follow-up time for progression was 10.3 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 35.0 [26.6 to 44.1]

3. Secondary Outcome: Overall Response Rate After at Least 12 Cycles of Treatment Assessed by the Independent Review Committee
Description: as for outcome 1
Time Frame: Response was assessed every 28 days until disease progression; ORR was analyzed after all participants received at least 12 cycles or discontinued treatment; the data cut-off date was 15 March 2019; median follow-up time for progression was 12.8 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 35.8 [27.3 to 44.9]

4. Secondary Outcome: Overall Response Rate After at Least 12 Cycles of Treatment Assessed by the Investigator
Description: as for outcome 1
Time Frame: Response was assessed every 28 days until disease progression; ORR was analyzed after all participants received at least 12 cycles or discontinued treatment; the data cut-off date was 15 March 2019; median follow-up time for progression was 13.1 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 35.0 [26.6 to 44.1]

5. Secondary Outcome: Clinical Benefit Rate After at Least 6 Cycles of Treatment Assessed by the Independent Review Committee
Description: Clinical benefit rate (CBR) is defined as the percentage of participants with the best overall response of minimal response (MR) or better according to International Myeloma Working Group Uniform Response Criteria (IMWG-URC) (i.e., a minimal response, partial response, very good partial response, complete response, or stringent complete response).
  MR: 25% to 49% reduction in the level of serum M-protein and a 50% to 89% reduction in 24-hour urinary M-protein, which still exceeds 200 mg /24 hour; If present at baseline, a >50% reduction in the size of soft tissue plasmacytomas is also required
Time Frame: Response was assessed every 28 days until disease progression; CBR was analyzed after all participants received at least 6 cycles or discontinued treatment; the data cut-off date was 05 November 2018; median follow-up time for progression was 8.9 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 48.0 [38.9 to 57.2]

6. Secondary Outcome: Clinical Benefit Rate After at Least 6 Cycles of Treatment Assessed by the Investigator
Description: Clinical benefit rate (CBR) is defined as the percentage of participants with the best overall response of minimal response (MR) or better according to IMWG-URC criteria (i.e., a minimal response, partial response, very good partial response, complete response, or stringent complete response).
  MR: 25% to 49% reduction in the level of serum M-protein and a 50% to 89% reduction in 24-hour urinary M-protein, which still exceeds 200 mg /24 hour; If present at baseline, a >50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: Response was assessed every 28 days until disease progression; CBR was analyzed after all participants received at least 6 cycles or discontinued treatment; the data cut-off date was 05 November 2018; median follow-up time for progression was 10.3 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 46.3 [37.3 to 55.6]

7. Secondary Outcome: Clinical Benefit Rate After at Least 12 Cycles of Treatment Assessed by the Independent Review Committee
Description: as for outcome 6
Time Frame: Response was assessed every 28 days until disease progression; CBR was analyzed after all participants received at least 12 cycles or discontinued treatment; the data cut-off date was 15 March 2019; median follow-up time for progression was 12.8 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 48.0 [38.9 to 57.2]

8. Secondary Outcome: Clinical Benefit Rate After at Least 12 Cycles of Treatment Assessed by the Investigator
Description: as for outcome 6
Time Frame: Response was assessed every 28 days until disease progression; CBR was analyzed after all participants received at least 12 cycles or discontinued treatment; the data cut-off date was 15 March 2019; median follow-up time for progression was 13.1 months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
percentage of participants | 46.3 [37.3 to 55.6]

9. Secondary Outcome: Duration of Overall Response (DOR)
Description: Duration of response (DOR) is defined as the time from first evidence of PR or better to disease progression (PD) or death due to any cause per the IMWG-URC criteria.
  PD:
  * Increase of 25% from lowest response value in any of the following:
    * Serum M-component (absolute increase ≥ 0.5 g/dL) and/or
    * Urine M-component (absolute increase ≥ 200 mg/24 hours)
    * In patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL)
  * Definite development of new or increase in size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcemia attributed solely to the plasma cell proliferative disorder.
  DOR was analyzed using the Kaplan-Meier method; Participants with no documented progression or death were censored at the date of their last disease assessment.
  DOR was determined based on both investigator and independent review committee response assessments.
Time Frame: Response was assessed every 28 days until disease progression; the data cut-off date was 15 March 2019; median follow-up time for progression assessed by independent review committee and by investigators were 12.8 months and 13.1 months, respectively.
Population: Safety population participants who achieved an overall response (best response of PR or better)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 44
months
  Independent Review Committee Assessment | 12.2 [7.4 to NA] — Could not be estimated due to the low number of events at the analysis cut-off date
  Investigator Assessment: number analyzed (Participants) | 43
  Investigator Assessment | 9.7 [7.4 to NA] — Could not be estimated due to the low number of events at the analysis cut-off date

10. Secondary Outcome: Duration of Clinical Benefit (DCB)
Description: Duration of clinical benefit (DCB) is defined as the time from first evidence of MR or better to disease progression or death due to any cause based on the (IMWG-URC criteria. DCB was estimated using the Kaplan-Meier method; participants with no disease progression or death at the analysis cut-off date were censored at their last disease assessment date.
  Duration of clinical benefit was determined based on both investigator and independent review committee response assessments.
Time Frame: as for outcome 9
Population: Safety population participants who achieved a best overall response of minimal response or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 59
months
  Independent Review Committee Assessment | 8.3 [7.3 to 15.1]
  Investigator Assessment: number analyzed (Participants) | 57
  Investigator Assessment | 8.6 [7.4 to 15.1]

11. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from first dose of any study treatment to the earlier of disease progression or death due to any cause according to the IMWG-URC criteria. PFS was analyzed using the Kaplan-Meier method; participants with no disease progression or death at the time of the data cut-off date were censored at the date of their last disease assessment; participants who started new anti-cancer therapy before disease progression or death were censored at their last disease assessment prior to starting new anti-cancer therapy.
  Progression-free survival was determined based on both investigator and independent review committee response assessments.
Time Frame: as for outcome 9
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
months
  Independent Review Committee Assessment | 5.6 [4.6 to 6.5]
  Investigator Assessment | 5.5 [4.6 to 6.5]

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the first dose of any study treatment to the date of death due to any cause. Overall survival was analyzed using the Kaplan-Meier method; participants who were alive or lost to follow-up as of the data analysis cut-off date were censored at their date of last contact (last known to be alive).
Time Frame: From first dose until the data cut-off date of 15 March 2019; median time on follow-up for survival was 15.3 months.
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 123
months | 15.2 [11.5 to NA] — Could not be estimated due to the low number of events at the time of the analysis.

13. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) is the time from the first dose of any study treatment to the first confirmed response (PR or better) based on both investigator and independent review committee response assessments.
Time Frame: as for outcome 9
Population: Safety population participants who achieved an overall response (best response of PR or better)
Measure: Median (Full Range); unit: months
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 44
months
  Independent Review Committee Assessment | 1.0 [1 to 11]
  Investigator Assessment: number analyzed (Participants) | 43
  Investigator Assessment | 1.0 [1 to 11]

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Carfilzomib
Description: Cmax is the maximum observed plasma concentration over the concentration-time profile of carfilzomib.
Time Frame: Cycles 1 and 2, day 1 at predose, 5 minutes after the start of carfilzomib infusion, immediately before the end of infusion, and at 5, 15, and 30 minutes, and 1, 2, and 4 hours after the end of infusion.
Population: Pharmacokinetic (PK) analyses were conducted on a subset of participants at selected sites. The PK analysis population included participants who received at least 1 dose of carfilzomib and had adequate data for the noncompartmental estimation of PK parameters. Results are reported for participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 24
ng/mL
  Cycle 1 Day 1 (20 mg/m²) | 744 (326)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 1210 (678)

15. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Carfilzomib
Description: Tmax of carfilzomib is the time at which maximum observed plasma concentrations of carfilzomib were observed.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 24
hours
  Cycle 1 Day 1 (20 mg/m²) | 0.50 [0.083 to 0.63]
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 0.50 [0.083 to 0.60]

16. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 to the Last Measurable Concentration (AUClast) for Carfilzomib
Description: AUClast of carfilzomib is the total area under the concentration-time curve beginning from time 0 to the time of the last measurable concentration of carfilzomib.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 24
hr*ng/mL
  Cycle 1 Day 1 (20 mg/m²) | 254 (102)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 401 (173)

17. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 Extrapolated to Infinity (AUC0-inf) for Carfilzomib
Description: AUC0-inf of carfilzomib is the total area under the concentration-time curve beginning from time 0 extrapolated to infinity following carfilzomib dosing.
Time Frame: as for outcome 14
Population: Pharmacokinetic analyses were conducted on a subset of participants at selected sites. Results are reported for participants in the PK analysis population with available data at each time point. PK profiles with a coefficient of determination (R²; goodness of fit) < 0.8 or percent extrapolated AUC > 20% were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 23
hr*ng/mL
  Cycle 1 Day 1 (20 mg/m²) | 256 (104)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 401 (173)

18. Secondary Outcome: Terminal Elimination Half-Life (T½) for Carfilzomib
Description: The terminal elimination half-life is the time required for plasma concentrations to fall by 50% in the terminal phase of the concentration-time profile.
Time Frame: as for outcome 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 23
hours
  Cycle 1 Day 1 (20 mg/m²) | 0.651 (0.259)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 0.792 (0.281)

19. Secondary Outcome: Systemic Clearance (CL) of Carfilzomib After Intravenous Infusion
Description: Systemic clearance is a measure of the ability of the body to eliminate drug, expressed in units of volume per time.
Time Frame: as for outcome 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 23
L/hr
  Cycle 1 Day 1 (20 mg/m²) | 157 (61.4)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 153 (112)

20. Secondary Outcome: Volume of Distribution (Varea) of Carfilzomib
Description: Volume of distribution is a pharmacokinetic parameter relating the amount of drug in the body to the concentration of drug in plasma.
Time Frame: as for outcome 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 23
Liters
  Cycle 1 Day 1 (20 mg/m²) | 148 (88.7)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 164 (102)

21. Secondary Outcome: Volume of Distribution at Steady State (Vss) for Carfilzomib
Description: Volume of distribution at steady-state is a pharmacokinetic parameter that relates the amount of drug in the body at steady-state to the concentration of drug in the plasma.
Time Frame: as for outcome 14
Population: PK analyses were conducted on a subset of participants at selected sites. Results are reported for participants in the PK analysis population with available data at each time point. PK profiles with a coefficient of determination < 0.8, percent extrapolated AUC > 20%, or negative values for Vss were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 22
liters
  Cycle 1 Day 1 (20 mg/m²) | 35.0 (20.2)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 27.2 (17.4)

22. Secondary Outcome: Mean Residence Time Observed From Time Zero to the Last Quantifiable Concentration (MRTlast) for Carfilzomib
Description: MRTlast is the mean residence time observed from time 0 until the time of the last quantifiable concentration.
Time Frame: as for outcome 14
Population: PK analyses were conducted on a subset of participants at selected sites. Results are reported for the participants in PK analysis population with available data at each time point. PK profiles with a coefficient of determination < 0.8, percent extrapolated AUC > 20%, or negative values for MRT were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Carfilzomib With Dexamethasone
Number analyzed (Participants) | 23
hours
  Cycle 1 Day 1 (20 mg/m²) | 0.225 (0.0856)
  Cycle 2 Day 1 (27 mg/m²): number analyzed (Participants) | 19
  Cycle 2 Day 1 (27 mg/m²) | 0.196 (0.0975)

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from the date enrolled until the end of study, median (minimum, maximum) time on study was 14.32 (0.066, 47.28) months. Adverse events are reported from the first dose of any study treatment up to 30 days after the end of study treatment, or initiation of new antimyeloma therapy, whichever occurred first; median (minimum, maximum) duration of treatment was 20.3 (0.3, 203) weeks.
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Carfilzomib With Dexamethasone
All-Cause Mortality (participants affected / at risk) | 91/126
Serious Adverse Events (participants affected / at risk) | 68/123
Other Adverse Events (participants affected / at risk) | 123/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib With Dexamethasone (N=123)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardiac amyloidosis (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 8
Disease progression (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 26
Respiratory tract infection (Infections and infestations) | 4
Soft tissue infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Myelopathy (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib With Dexamethasone (N=123)
Anaemia (Blood and lymphatic system disorders) | 76
Leukocytosis (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Vision blurred (Eye disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 8
Oedema peripheral (General disorders) | 12
Peripheral swelling (General disorders) | 9
Pyrexia (General disorders) | 22
Hepatic function abnormal (Hepatobiliary disorders) | 7
Bronchitis (Infections and infestations) | 12
Influenza (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 28
Respiratory tract infection (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 60
Alanine aminotransferase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 12
Bilirubin conjugated increased (Investigations) | 9
Blood albumin decreased (Investigations) | 10
Blood bilirubin increased (Investigations) | 17
Blood creatinine increased (Investigations) | 23
Blood glucose increased (Investigations) | 17
Blood lactate dehydrogenase increased (Investigations) | 20
Blood phosphorus increased (Investigations) | 10
Blood potassium decreased (Investigations) | 12
Blood pressure increased (Investigations) | 18
Blood urea increased (Investigations) | 15
Blood uric acid increased (Investigations) | 18
Gamma-glutamyltransferase increased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 34
Lymphocyte percentage decreased (Investigations) | 12
Mean cell volume increased (Investigations) | 8
Neutrophil count decreased (Investigations) | 37
Neutrophil count increased (Investigations) | 20
Neutrophil percentage increased (Investigations) | 15
Platelet count decreased (Investigations) | 60
Prealbumin decreased (Investigations) | 9
White blood cell count decreased (Investigations) | 48
White blood cell count increased (Investigations) | 17
Hypercalcaemia (Metabolism and nutrition disorders) | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 21
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 20
Hypokalaemia (Metabolism and nutrition disorders) | 43
Hyponatraemia (Metabolism and nutrition disorders) | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Hypoproteinaemia (Metabolism and nutrition disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 9
Neuropathy peripheral (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12
Hypertension (Vascular disorders) | 47
Hypoglycaemia (Metabolism and nutrition disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT03029234/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03029234/SAP_001.pdf